CLINICAL TRIAL: NCT04983628
Title: Prognostic and Predictive Value of Tumor Molecular Alterations in Patients With Prostate Cancer
Brief Title: Molecular Profiling in Prostate Cancer
Acronym: ProProstate
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: TR_9/21
Record Dates: First submitted 2021-02-16; First posted 2021-07-30 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer Metastatic; Prostate Cancer Recurrent; Germline BRCA1 Gene Mutation; Germline BRCA2 Gene Mutation; Mutation
Keywords: Prostate cancer; Predictive biomarker; Prognostic biomarker
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Formalin-fixed paraffin-embedded tissue samples and germline DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tumor molecular profiling — targeted DNA NGS

SUMMARY:
We aim to employ targeted DNA NGS to evaluate the prevalence of germline and somatic mutations in cancer predisposing genes, such as BRCA1 and BRCA2, and other HR and DDR genes, including also a few additional clinically relevant genes, in patients with metastatic, locally advanced or high-grade prostate cancer. In addition, we will investigate the prognostic role of these mutations as well as their association with various clinicopathological parameters. This will be the first study investigating the prevalence of germline and somatic pathogenic mutations in Greek patients with prostate cancer.

DETAILED DESCRIPTION:
This study will include formalin-fixed paraffin-embedded tumor tissue (FFPE) from 250 patients with metastatic, recurrent, locally advanced or "intermediate or high risk" (Gleason >7), operable prostate cancer. FFPE tumor blocks alongside peripheral blood will be retrieved for all patients from Pathology Laboratories. Available FFPE blocks will be subjected to histological review by an experienced pathologist to evaluate H&E sections for confirmation of diagnosis, histologic type, grade and tumor cell content (TCC%), as well as mark tumor dense areas for manual macro-dissection, prior to DNA extraction, in order to enrich samples for tumor DNA. Clinicopathologic characteristics of patients with prostate cancer will be retrieved from their respective medical records. Diagnosis will be confirmed through pathology reports, which will also provide information about Gleason Score and histological subtype.

In all instances, the collection of patient information will be in compliance with the regulations of the Bioethics committees of participating Hospitals. The study will be conducted in accordance with the principles of the Helsinki Declaration of Human Rights.

Following manual macro-dissection, FFPE tumor tissue material will be processed for DNA extraction, according to standard procedures with the QIAamp DNA Mini Kit (Qiagen GmbH, Hilden, Germany).

Sequencing will be performed at the Laboratory of Molecular Oncology, using an Ion Torrent Proton Sequencer (Life Technologies/Ion Torrent). For the purpose of targeted NGS genotyping of tumor and available matched germline DNA samples, we designed a custom Ampliseq panel to target coding relevant regions of genes involved in homologous recombination (HR), along with several others.

Data retrieval and base calling will be performed on the Torrent Server (v5.8.0.8). Consequently, we will then employ appropriate Ion Reporter Workflows (version 5.10) to automatically annotate single nucleotide variants (SNVs), multiple nucleotide variants (MNVs), small insertions / deletions (INDELs) and copy number variations (CNVs).

ELIGIBILITY:
Inclusion Criteria:

* metastatic prostate cancer
* recurrent prostate cancer
* locally advanced prostate cancer
* "intermediate or high risk" (Gleason >7), operable prostate cancer
* available FFPE tumor tissue

Exclusion Criteria:

* absence of tumor tissue available for analysis

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with metastatic, recurrent, locally advanced or "intermediate or high risk" (Gleason >7), operable prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of germline and somatic mutations in cancer predisposing genes | 1 year
  Number of patients with either germline or somatic mutations

SECONDARY OUTCOMES:
Overall survival | 3 years
  Time from diagnosis to the date of death, through the completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Elena Fountzila, Principal Investigator — HeCOG
Locations (1):
- Hellenic Cooperative Oncology Group, Athens, Greece

IPD SHARING:
Plan to Share IPD: No